CLINICAL TRIAL: NCT05516108
Title: Smartphone-based Mindfulness Training for Health Following Early Life Adversity
Brief Title: Remote Mindfulness Training Following Early Life Adversity
Acronym: ReMind
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Emily Lindsay, Research Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY21030189; K01AT011232 (NIH)
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Stress; Mindfulness; Early Life Adversity
MeSH Terms: interventions — Mindfulness; Coping Skills

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): Mindfulness intervention involving 14 foundational audio-guided lessons plus daily brief practice prompts. Lessons train meditation techniques for 3 mindfulness skills: concentration, sensory clarity, and equanimity. Practice prompts delivered 3x daily build on the skills trained in each lesson.
  Interventions: Behavioral: Mindfulness
- Coping (Active Comparator): Coping intervention involving 14 foundational audio-guided lessons plus daily brief practice prompts. Lessons train techniques for 3 coping skills: reflection, reappraisal, and problem solving. Practice prompts delivered 3x daily build on the skills trained in each lesson.
  Interventions: Behavioral: Coping

INTERVENTIONS:
Behavioral: Mindfulness — The mindfulness intervention includes 14 daily 20-minute audio lessons plus brief daily practice prompts. Lessons train specific meditation techniques through didactic explanation and guided practice. Based on the Unified Mindfulness system, lessons train 3 mindfulness skills: concentration, sensory clarity, and equanimity. Concentration, a state of stable attention on the intended target, enables participants to monitor present-moment physical and emotional body experiences. Sensory clarity, the monitoring of momentary experiences, involves detecting subtle sensations and discriminating between different experiences. Equanimity, an attitude of acceptance toward momentary experiences, is trained through 3 strategies: (a) body relaxation, (b) mental welcoming, and (c) a gentle tone of voice. Practice prompts build on the skills trained in each lesson, encouraging participants to practice brief moments of mindful awareness, mindfulness while doing daily tasks, or formal meditation.
  Arms: Mindfulness
Behavioral: Coping — The coping intervention includes 14 daily 20-minute audio lessons plus brief daily practice prompts. Lessons train specific coping techniques through didactic explanation and guided practice. Lessons train coping skills (reflection, reappraisal, and problem solving) without encouraging focus on or acceptance of present experience (i.e., mindfulness skills). Participants are instructed to: (1) reflect and let their minds drift, (2) reframe or reappraise past and anticipated events, and (3) analyze and solve personal problems. Practice prompts build on the skills trained in each lesson, encouraging participants to take brief reflection breaks or to practice reappraisal or problem-solving skills.
  Arms: Coping

SUMMARY:
This study will test the feasibility of delivering smartphone-based mindfulness and coping interventions to a sample of emerging/young adults with a history of early life adversity (ELA). 80 participants with a history of ELA will be randomly assigned to complete a two-week mindfulness training intervention or matched coping control intervention, both involving 14 foundational audio-guided lessons and practice prompts randomly delivered 3x daily. At baseline, post-intervention, and one-month follow-up lab assessments, participants will complete questionnaires and provide blood samples for assessment of markers of inflammation. Data assessing subjective and physiological stress in daily life will be collected during the intervention and for one week before, immediately after, and one month after the intervention. Passive sensor data will be continuously collected from participants' smartphones and wearable devices to develop exploratory models that estimate and predict daily life stress. Data will be used to evaluate feasibility and acceptability of interventions and assessments in an ELA sample, test effects of mindfulness training on daily life stress and markers of inflammation in an ELA sample, and develop exploratory machine learning models of stress from passive sensor data.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-29 years
* English speaking
* History of moderate-to-severe physical, emotional, or sexual abuse in childhood
* Data-enabled Android or iOS smartphone
* Able to meet study requirements

Exclusion Criteria:

* Self-reported diagnosis of chronic physical disease (e.g., cancer, HIV, heart disease, diabetes, bleeding disorder)
* Self-reported diagnosis of chronic mental disorder (e.g., schizophrenia, personality disorder, or psychotic illness), major neurological disorder, or suicidal thoughts or wishes at baseline
* Substance use disorder
* Medication use that interferes with HPA-axis activity (e.g., corticosteroids), autonomic activity (e.g., antihypertensive medication), inflammatory activity (e.g., cholesterol medications), or blood clotting
* Current antibiotic, antiviral, or antimicrobial treatment
* Shift workers
* Pregnancy
* Regular systematic mind-body practice (>2 times per week)

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K Lindsay, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All data sharing will follow NIH and Pitt IRB guidelines. To gain access to IPD that underlie results in a publication, anyone not part of the original research will submit a Data Analysis Request Form, which requires a description of hypotheses, specific data requested, and investigator information. The investigator must complete the Pitt Certification Program in Research Practice Fundamentals or a comparable program. Upon approval, a de-identified dataset and codebook will be provided. Investigators outside Pitt must also complete a Data Use and Confidentiality Agreement. This signed letter of agreement states that the investigator (1) will cite the original study dataset and funding source in all presentations and publications, and (2) will not share these data and study materials with others. Participants will be made aware of the potential for sharing of de-identified data with outside investigators on informed consent documents.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Upon request, data collected for this study will also be made available to other investigators following publication of primary findings.
Access Criteria: Data Analysis Request Form; completion of the University of Pittsburgh Certification Program in Research Practice Fundamentals or a comparable training program at their own institution; Data Use and Confidentiality Agreement for investigators outside University of Pittsburgh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited into this study between August 2022 and March 2024. The study was advertised through "Pitt+Me," a registry of over 300,000 individuals in the Pittsburgh area interested in participating in research.
Period: Overall Study
Arm/Group | Mindfulness | Coping
Started | 42 | 39
Completed | 37 | 34
Not Completed | 5 | 5
Not completed — Time Commitment | 3 | 1
Not completed — Reason Unknown | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness | Coping | Total
Number analyzed (Participants) | 42 | 39 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.02 (3.11) | 23.79 (3.50) | 23.91 (3.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 36 | 69
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 39 | 37 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 8 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 18 | 21 | 39
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 42 | 39 | 81

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment (Screened Eligible)
Description: Recruitment benchmark: >10% of people screened will be eligible
Time Frame: assessed pre-enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Screening & Enrollment: All individuals who were pre-screened for eligibility before randomization.
Arm/Group | Screening & Enrollment
Number analyzed (Participants) | 891
Participants
  Screened eligible at in-person screening | 81
  Pre-screened eligible but screened ineligible at in-person screening | 56
  Pre-screened eligible but did not attend in-person screening | 112
  Pre-screened ineligible | 642

2. Primary Outcome: Feasibility of Retention
Description: Retention benchmark: >80% retention through intervention and >75% retention through follow-up
Time Frame: assessed across the entire 8-week study period
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
Participants
  Retained through follow-up assessments | 37 | 34
  Did not complete intervention | 4 | 5
  Completed intervention but did not complete follow-up assessments | 1 | 0

3. Primary Outcome: Feasibility of Adherence: Intervention Lessons
Description: Numbers represent percentages of intervention lessons completed in mindfulness and coping groups [calculated as (average number of lessons completed / 14 total lessons among all participants in each group) * 100]. The original adherence benchmark was an average completion of >85% of intervention lessons; reported percentages that are greater than that benchmark represent feasibility of intervention adherence.
Time Frame: assessed across the entire 2-week intervention period
Population: study completers
Measure: Number; unit: percentage of lessons completed
Units Other Than Participants: intervention lessons
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 37 | 34
Number analyzed (intervention lessons) | 14 | 14
percentage of lessons completed | 94.57 | 94.71

4. Primary Outcome: Feasibility of Safe Implementation: Incidence of Treatment-emergent Increases in Mental Health Symptoms
Description: Safety benchmark: <10% of participants showing substantial (>2SD) increases in anxiety, trauma, or depressive symptoms (using PROMIS Anxiety and Depression scales and Posttraumatic Stress Disorder Checklist-Civilian scale described in other outcomes below) combined to create treatment-emergent symptom rate
Time Frame: assessed across the entire 8-week study period
Population: intervention completers
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 38 | 34
Participants
  No substantial (>2SD) symptom increase | 35 | 34
  Substantial (>2SD) symptom increase at post-intervention or follow-up | 3 | 0

5. Primary Outcome: Acceptability: Treatment Expectancies
Description: Acceptability of interventions, with benchmark of >80% of participants giving positive ratings of treatment expectancies (>3 on 6-item Credibility/Expectancy Questionnaire)
Time Frame: assessed in-person at post-intervention laboratory assessment (an average of 4 weeks) and one-month follow-up laboratory assessment (an average of 8 weeks)
Population: study completers
Measure: Number; unit: percentage of treatment completers
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 37 | 34
percentage of treatment completers
  Post-intervention | 95 | 91
  One-month follow-up | 92 | 88

6. Primary Outcome: Change in Daily Life Subjective Stress: State Perceived Stress
Description: State perceived stress assessed in daily life four times per day for one week at three time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Stress was assessed on a 1-7 Likert scale, with higher scores indicating higher perceived stress.
Time Frame: change in stress assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
units on a scale
  Pre-intervention | 2.48 (.13) | 2.5 (.13)
  Post-intervention | 2.56 (.13) | 2.37 (.13)
  One-month follow-up | 2.46 (.13) | 2.32 (.13)
Statistical Analysis 1: Comparison: Mindfulness vs Coping; time (pre, post, follow-up) x condition (mindfulness, coping); Test type: Other; p = .004, Mixed Models Analysis; Stata mixed

7. Primary Outcome: Change in Daily Life Subjective Stress: Daily Perceived Stress
Description: Daily perceived stress assessed in daily life each evening for one week at three time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Stress was assessed on a 1-7 Likert scale, with higher scores indicating higher perceived stress.
Time Frame: as for outcome 6
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
units on a scale
  Pre-intervention | 3.01 (.14) | 2.91 (.15)
  Post-intervention | 3.19 (.15) | 2.69 (.15)
  One-month follow-up | 2.90 (.15) | 2.63 (.15)
Statistical Analysis 1: Comparison: Mindfulness vs Coping; time (pre, post, follow-up) x condition (mindfulness, coping); Test type: Other; p = .020, Mixed Models Analysis

8. Primary Outcome: Change in Daily Life Objective Stress: Stress Events in the Past 2.5 Hours
Description: Stress events assessed on a binary scale (yes/no) in daily life four times per day for one week at three time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in logistic MLM analyses. Outcomes are reported as mean percentage of surveys at each time point that stress events were endorsed, with higher percentages indicating more stress events.
Time Frame: as for outcome 6
Measure: Mean (Standard Error); unit: percentage of surveys with stressors
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
percentage of surveys with stressors
  Pre-intervention | 22.71 (2.26) | 18.5 (2.09)
  Post-intervention | 15.84 (1.91) | 12.33 (1.72)
  One-month follow-up | 15.31 (1.89) | 10.78 (1.6)
Statistical Analysis 1: Comparison: Mindfulness vs Coping; time (pre, post, follow-up) x condition (mindfulness, coping); Test type: Other; p = .74, Mixed Models Analysis; Stata melogit

9. Primary Outcome: Change in Daily Life Objective Stress: Daily Stress Events
Description: Daily stress events assessed in daily life each evening for one week at three time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in logistic MLM analyses. Outcomes are reported as mean percentage of days at each time point that stress events were endorsed, with higher percentages indicating more stress events.
Time Frame: as for outcome 6
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: percentage of days with stressors
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
percentage of days with stressors
  Pre-intervention | 65.93 (4.01) | 51.52 (4.46)
  Post-intervention | 57.54 (4.46) | 47.75 (4.69)
  One-month follow-up | 48.18 (4.61) | 46.08 (4.70)
Statistical Analysis 1: Comparison: Mindfulness vs Coping; time (pre, post, follow-up) x condition (mindfulness, coping); Test type: Other; p = .10, Mixed Models Analysis

10. Primary Outcome: Change in Daily Life Physiological Stress Reactivity
Description: Heart Rate (HR) measured continuously in daily life, with HR averaged in 30-minute windows around daily life stress reported via EMA up to four times per day for one week at three time points, totaling up to 28 windows at each time point. All (up to) 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher scores indicate higher HR in beats per minute (relative to an individual's average daily HR) at high stress moments (relative to an individual's average perceived stress).
Time Frame: change in HR reactivity assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Population: all available data; n=5 participants provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 39 | 37
beats per minute
  Pre-intervention | 5.82 (.67) | 4.77 (.68)
  Post-intervention | 4.94 (.69) | 6.49 (.73)
  One-month follow-up | 6.6 (.73) | 5.80 (.78)
Statistical Analysis 1: Comparison: Mindfulness vs Coping; time (pre, post, follow-up) x condition (mindfulness, coping); Test type: Other; p = .009, Mixed Models Analysis; Stata mixed

11. Primary Outcome: Change in Circulating Inflammatory Markers
Description: Circulating IL-6 assessed via dried blood spot (DBS), reported as raw concentration in pg/mL assessed via ProteinSimple Simple Plex Human IL-6 (3rd gen) on Ella instrument
Time Frame: change from pre-intervention laboratory assessment to post-intervention laboratory assessment (an average of 4 weeks) and one-month follow-up laboratory assessment (an average of 8 weeks)
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
pg/mL
  pre-intervention | .365 (.034) | .266 (.035)
  post-intervention | .343 (.036) | .267 (.038)
  one-month follow-up | .344 (.036) | .279 (.037)

12. Primary Outcome: Feasibility of Recruitment (Enrollment)
Description: Recruitment benchmark: >60% of those eligible will enroll
Time Frame: assessed pre-enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Screening & Enrollment
Number analyzed (Participants) | 81
Participants | 81

13. Primary Outcome: Feasibility of Adherence: Intervention Practice Prompts
Description: Numbers represent percentages of intervention practice prompts completed in mindfulness and coping groups [calculated as (average number of prompts completed / 42 total prompts among all participants in each group) * 100]. The original adherence benchmark was an average completion of >60% of prompts; reported percentages that are greater than that benchmark represent feasibility of intervention practice prompt adherence.
Time Frame: assessed across the entire 2-week intervention period
Population: study completers
Measure: Number; unit: percentage of prompts completed
Units Other Than Participants: intervention practice prompts
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 37 | 34
Number analyzed (intervention practice prompts) | 42 | 42
percentage of prompts completed | 57.33 | 60.34

14. Primary Outcome: Feasibility of Adherence: Ambulatory Assessments
Description: Numbers represent percentages of ambulatory assessment surveys completed in mindfulness and coping groups [calculated as (average number of surveys completed / 105 total surveys among all participants in each group) * 100]. The original adherence benchmark was an average completion of >75% of ambulatory assessments; reported percentages that are greater than that benchmark represent feasibility of ambulatory assessment adherence.
Time Frame: assessed for 1 week at three time points: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Population: study completers
Measure: Number; unit: percentage of surveys completed
Units Other Than Participants: ambulatory assessment surveys
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 37 | 34
Number analyzed (ambulatory assessment surveys) | 105 | 105
percentage of surveys completed | 86.28 | 87.53

15. Primary Outcome: Feasibility of Adherence: Mobile Sensor Data
Description: Numbers represent percentages of days on which wearable sensor (Fitbit) data and AWARE phone sensor data were collected in mindfulness and coping groups [calculated as (average number of days that Fitbit/AWARE data were collected / 56 days among all participants in each group) * 100]. The original adherence benchmark was collecting mobile sensor data on >75% of days; reported percentages that are greater than that benchmark represent feasibility of mobile sensor data collection adherence.
Time Frame: assessed across the entire 8-week study period
Population: study completers
Measure: Number; unit: percentage of days
Units Other Than Participants: days of mobile sensor data collection
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 37 | 34
Number analyzed (days of mobile sensor data collection) | 56 | 56
percentage of days
  % of days Fitbit data collected | 86.95 | 86.40
  % of days AWARE data collected | 94.35 | 91.61

16. Secondary Outcome: Change in Daily Life Positive Affect: State
Description: State positive affect assessed in daily life four times per day for one week at three time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Positive affect was assessed on a 1-7 Likert scale, with higher scores indicating higher positive affect.
Time Frame: change in affect assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
units on a scale
  Pre-intervention | 3.87 (.14) | 3.77 (.14)
  Post-intervention | 3.57 (.14) | 3.80 (.14)
  One-month follow-up | 3.74 (.14) | 3.75 (.14)

17. Secondary Outcome: Change in Daily Life Positive Affect: Daily
Description: Daily positive affect (composite of 9 positive affect items across 3 subscales: happiness (happy, pleased, and cheerful), calm (calm, at-ease, and relaxed), and vigor (lively, full-of-pep, and energetic), each assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at three time points via end-of day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher scores reflect higher positive affect.
Time Frame: as for outcome 16
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
units on a scale
  Pre-intervention | 3.30 (.14) | 3.34 (.14)
  Post-intervention | 2.94 (.14) | 3.32 (.15)
  One-month follow-up | 3.19 (.14) | 3.36 (.15)

18. Secondary Outcome: Change in Daily Life Negative Affect: State
Description: State negative affect assessed in daily life four times per day for one week at three time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Negative affect was assessed on a 1-7 Likert scale, with higher scores indicating higher negative affect.
Time Frame: as for outcome 16
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
units on a scale
  Pre-intervention | 2.19 (.11) | 2.06 (.12)
  Post-intervention | 2.34 (.11) | 1.96 (.12)
  One-month follow-up | 2.21 (.11) | 1.93 (.12)

19. Secondary Outcome: Change in Daily Life Negative Affect: Daily
Description: Daily negative affect (composite of 9 negative affect items across 3 subscales: anxiety (on edge, nervous, and tense), depression (sad, depressed, and unhappy), and hostility (hostile, resentful, and angry), each assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at three time points via end-of day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher scores reflect higher negative affect.
Time Frame: as for outcome 16
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
units on a scale
  Pre-intervention | 2.15 (.11) | 1.99 (.11)
  Post-intervention | 2.19 (.11) | 1.88 (.11)
  One-month follow-up | 2.13 (.11) | 1.82 (.11)

20. Secondary Outcome: Change in Daily Life Social Interactions: Interactions in the Past 2.5 Hours
Description: Number of social interactions assessed in daily life four times per day for one week at three time points via Ecological Momentary Assessment (EMA), totaling up to 28 assessments at each time point. All 28 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher numbers indicate more social interactions.
Time Frame: change in interactions assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Measure: Mean (Standard Error); unit: number of interactions
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
number of interactions
  Pre-intervention | 2.79 (.26) | 2.96 (.27)
  Post-intervention | 3.09 (.26) | 2.84 (.27)
  One-month follow-up | 3.30 (.26) | 2.69 (.27)

21. Secondary Outcome: Change in Daily Life Social Interactions: Daily
Description: Number of social interactions assessed in daily life each evening for one week at three time points via end-of day diary, totaling up to 7 assessments at each time point. All 7 assessments at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher numbers indicate more social interactions.
Time Frame: as for outcome 20
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: number of interactions
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
number of interactions
  Pre-intervention | 12.69 (.78) | 11.59 (.80)
  Post-intervention | 13.60 (.79) | 11.18 (.82)
  One-month follow-up | 14.61 (.80) | 11.25 (.82)

22. Secondary Outcome: Change in Daily Life Mindfulness: Awareness
Description: Mindful awareness (composite 3-item scale: "Today, I paid attention to what I was doing in the present moment" / "Today, I noticed body sensations come and go" / "Today, I noticed pleasant and unpleasant thoughts and emotions", each item assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at three time points via end-of-day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher composite scores reflect higher mindful awareness.
Time Frame: change in awareness assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
score on a scale
  Pre-intervention | 3.76 (.15) | 3.70 (.16)
  Post-intervention | 3.98 (.16) | 4.10 (.16)
  One-month follow-up | 4.03 (.16) | 4.10 (.16)

23. Secondary Outcome: Change in Daily Life Mindfulness: Acceptance
Description: Mindful acceptance (composite 2-item scale: "Today, I was able to step back and be aware of distressing thoughts, emotions, and sensations, without being taken over by them" / "Today, I did not want to feel the way I was feeling", each item assessed on a 1-7 Likert scale) assessed in daily life each evening for one week at three time points via end-of-day diary, totaling up to 7 scores at each time point. All 7 composite scores at each of the three time points (pre-intervention ambulatory assessment, post-intervention ambulatory assessment, and one-month follow-up ambulatory assessment) were averaged in MLM analyses. Higher composite scores reflect higher acceptance.
Time Frame: change in acceptance assessed in daily life for 1 week at three timepoints: pre-intervention ambulatory assessment, post-intervention ambulatory assessment (an average of 3 weeks), and one-month follow-up ambulatory assessment (an average of 7 weeks)
Population: all available data; n=1 participant provided no data at pre-intervention, post-intervention, or follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 41 | 39
score on a scale
  Pre-intervention | 4.25 (.14) | 4.35 (.14)
  Post-intervention | 4.33 (.14) | 4.74 (.15)
  One-month follow-up | 4.63 (.14) | 4.82 (.15)

24. Other Pre Specified Outcome: Passive Sensor Stress Models
Description: Passive sensor data from smartphones (location, activity, screen status, battery, weather, time zone, communication) and wearable devices (heart rate, activity, sleep) combined to develop machine learning models predicting state stress
Time Frame: collected continuously for 8 weeks
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in State Stress Following Intervention Practice
Description: State stress following intervention practice used to evaluate immediate benefit of practice delivered at high-stress moments
Time Frame: change from pre- to post-practice across two-week intervention period
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Daily Stress Following Intervention Practice
Description: End-of-day stress on days with intervention practice used to evaluate day-level benefit of practice delivered at high-stress moments
Time Frame: daily stress across two-week intervention period
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Early Life Adversity: Childhood Trauma
Description: Assessed via the Childhood Trauma Questionnaire (a 28-item scale with three 5-item abuse subscales - physical, sexual, and emotional abuse - ranging from 5-25, with higher scores indicating higher childhood trauma)
Time Frame: pre-intervention
Measure: Mean (Standard Error); unit: CTQ score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
CTQ score
  Emotional abuse score | 14.76 (0.61) | 13.56 (0.64)
  Physical abuse score | 8.07 (0.57) | 7.72 (0.59)
  Sexual abuse score | 6.88 (0.60) | 7.10 (0.62)

28. Other Pre Specified Outcome: Early Life Adversity: Emotional Neglect
Description: Early Life Adversity assessed via the Childhood Experiences of Care and Abuse Inventory (a 16-item scale referencing mother and father figures, with an 8-item emotional neglect subscale ranging from 8-40, where higher scores indicate higher levels of emotional neglect)
Time Frame: pre-intervention
Measure: Mean (Standard Error); unit: CECA-Q score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
CECA-Q score
  Mother figure neglect | 13.67 (1.04) | 10.51 (1.08)
  Father figure neglect | 18.12 (1.20) | 17.15 (1.25)

29. Other Pre Specified Outcome: Early Life Adversity: Childhood SES Indexed Via Parental Education
Description: Childhood SES indexed via parental educational attainment, ranging from less than high school education to doctoral degree (1 = No High School Diploma, 2 = GED, 3 = High School Diploma, 4 = Technical Training, 5 = Some College, no degree, 6 = Associate Degree, 7 = Bachelor's Degree, 8 = Master's Degree, 9 = MD, PhD, JD, or PharmD), with higher scores indicating higher educational attainment
Time Frame: pre-intervention
Measure: Mean (Standard Error); unit: SES Score (Parental Education)
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
SES Score (Parental Education)
  Maternal education | 6.12 (0.32) | 6.46 (0.33)
  Paternal education | 5.95 (0.35) | 5.95 (0.37)

30. Other Pre Specified Outcome: Early Life Adversity: Childhood SES Indexed by Government Food Assistance
Description: Childhood SES assessed via National Comorbidity Survey: Adolescents item assessing government food assistance
Time Frame: pre-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
Participants | 14 | 11

31. Other Pre Specified Outcome: Early Life Adversity: Domestic Violence
Description: Early Life Adversity assessed via Adverse Childhood Experiences Survey (using a 5-item domestic violence subscale, ranging from 0-10, with higher scores indicating higher levels of domestic violence)
Time Frame: pre-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
Participants
  ACES criminal behavior | 1 | 4
  ACES domestic violence | 10 | 5

32. Other Pre Specified Outcome: Change in Circulating Inflammatory Biomarkers: CRP
Description: Circulating CRP assessed via dried blood spot (DBS) [additional funding needed to assess]
Time Frame: change from pre-intervention to post-intervention (an average of 4 weeks) and one-month follow-up (an average of 8 weeks)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change in Circulating Inflammatory Biomarkers: TNF
Description: Circulating TNF assessed via dried blood spot (DBS) [additional funding needed to assess]
Time Frame: as for outcome 32
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Change in Circulating Inflammatory Biomarkers: IL-8
Description: Circulating IL-8 assessed via dried blood spot (DBS) [additional funding needed to assess]
Time Frame: as for outcome 32
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Circulating Inflammatory Biomarkers: IL-10
Description: Circulating IL-10 assessed via dried blood spot (DBS) [additional funding needed to assess]
Time Frame: as for outcome 32
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Anxiety
Description: Assessed in-person via PROMIS Anxiety, a 4-item scale with raw scores ranging from 4-20 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher anxiety
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Anxiety Score (Pre-Intervention) | 61.37 (1.13) | 60.29 (1.17)
  Mean Anxiety Score (Post-Intervention) | 58.97 (1.16) | 56.99 (1.22)
  Mean Anxiety Score (1 Month Follow Up) | 58.56 (1.17) | 56.94 (1.22)

37. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Depressive Symptoms
Description: Assessed in-person via PROMIS Depression, a 4-item scale with raw scores ranging from 4-20 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher depressive symptoms
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Depressive Score (Pre-Intervention) | 56.90 (1.29) | 53.76 (1.34)
  Mean Depressive Score (Post-Intervention) | 55.76 (1.35) | 50.54 (1.42)
  Mean Depressive Score (1 Month Follow Up) | 55.86 (1.39) | 52.39 (1.45)

38. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Social Isolation
Description: Assessed in-person via PROMIS Social Isolation, a 14-item scale with raw scores ranging from 14 to 70 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher social isolation
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Social Isolation Score (Pre-Intervention) | 53.64 (1.42) | 50.55 (1.48)
  Mean Social Isolation Score (Post-Intervention) | 51.52 (1.45) | 49.64 (1.52)
  Mean Social Isolation Score (1 Month Follow Up) | 51.29 (1.46) | 48.80 (1.52)

39. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Perceived Stress
Description: Assessed in-person via Perceived Stress Scale (a 10-item scale ranging from 0-40, with higher scores indicating higher perceived stress)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean PSS Score (Pre-Intervention) | 21.60 (0.91) | 20.85 (0.94)
  Mean PSS Score (Post-Intervention) | 20.42 (0.96) | 16.92 (1.01)
  Mean PSS Score (1-Month Follow-Up) | 18.21 (0.99) | 16.81 (1.04)

40. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Trauma Symptoms
Description: Assessed in-person via Post-Traumatic Stress Disorder Checklist for Civilians (PCL-C), a 17-item scale ranging from 17-85, with higher scores indicating higher levels of trauma, and scores of 30 or greater indicating at least moderately severe PTSD symptoms
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean PCL Score (Pre-Intervention) | 40.19 (1.89) | 40.21 (1.97)
  Mean PCL Score (Post-Intervention) | 35.76 (1.95) | 31.44 (2.04)
  Mean PCL Score (1 Month Follow Up) | 34.63 (1.96) | 32.18 (2.04)

41. Other Pre Specified Outcome: Change in Global Psychosocial Stress: Depersonalization
Description: Assessed in-person via Cambridge Depersonalization Scale (a 29-item scale ranging from 0-116, assessing frequency and duration of depersonalization symptoms, with higher scores indicating greater depersonalization)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean CDS Score (Pre-Intervention) | 58.31 (6.02) | 52.15 (6.25)
  Mean CDS Score (Post-Intervention) | 47.49 (6.16) | 36.30 (6.45)
  Mean CDS Score (1 Month Follow Up) | 43.94 (6.19) | 30.83 (6.45)

42. Other Pre Specified Outcome: Change in Sleep Quality
Description: Assessed in-person via Pittsburgh Sleep Quality Index (6-item short form, ranging from 0-12, with higher scores indicating worse sleep)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean PSQI Score (Pre-Intervention) | 4.14 (0.37) | 4.28 (0.38)
  Mean PSQI Score (Post-Intervention) | 4.13 (0.33) | 3.20 (0.35)
  Mean PSQI Score (1 Month Follow Up) | 3.81 (0.34) | 3.85 (0.35)

43. Other Pre Specified Outcome: Change in Global Psychosocial Resilience: Life Satisfaction
Description: Assessed in-person via PROMIS Life Satisfaction, a 5-item scale with raw scores ranging from 5-35 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher life satisfaction
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Life Satisfaction Score (Pre-Intervention) | 41.47 (1.30) | 45.34 (1.35)
  Mean Life Satisfaction Score (Post-Intervention) | 42.35 (1.42) | 46.92 (1.49)
  Mean Life Satisfaction Score (1 Month Follow Up) | 43.79 (1.59) | 48.24 (1.65)

44. Other Pre Specified Outcome: Change in Global Psychosocial Resilience: Positive Affect
Description: Assessed in-person via PROMIS Positive Affect, a 15-item scale with raw scores ranging from 15-75 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher positive affect
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Positive Affect Score (Pre-Intervention) | 41.09 (1.17) | 44.16 (1.22)
  Mean Positive Affect Score (Post-Intervention) | 41.96 (1.24) | 45.15 (1.30)
  Mean Positive Affect Score (1 Month Follow Up) | 42.53 (1.28) | 44.16 (1.34)

45. Other Pre Specified Outcome: Change in Global Psychosocial Resilience: Self-Efficacy
Description: Assessed in-person via PROMIS Self-Efficacy, a 4-item scale with raw scores ranging from 4-20 and converted to t-scores, with t-scores of 50 (standard deviation = 10) representing the average for the US general population and higher t-scores indicating higher self-efficacy
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
t-score
  Mean Self-efficacy Score (Pre-Intervention) | 44.60 (1.47) | 45.32 (1.53)
  Mean Self-efficacy Score (Post-Intervention) | 45.73 (1.52) | 47.40 (1.59)
  Mean Self-efficacy Score (1 Month Follow Up) | 48.22 (1.53) | 47.55 (1.59)

46. Other Pre Specified Outcome: Change in Global Mindfulness
Description: Five Facet Mindfulness Questionnaire-Short Form (a 24-item scale including five subscales - observing, describing, acting with awareness, nonreactivity, and nonjudgment, with average scores ranging from 1-5 and higher scores indicating higher mindfulness)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean Global Mindfulness Score (Pre-Intervention) | 3.10 (0.07) | 3.15 (0.08)
  Mean Global Mindfulness Score (Post-Intervention) | 3.27 (0.08) | 3.44 (0.09)
  Mean Global Mindfulness Score (1 Month Follow Up) | 3.39 (0.09) | 3.49 (0.10)

47. Other Pre Specified Outcome: Change in Global Experiential Avoidance
Description: Acceptance and Action Questionnaire-II (a 7-item scale ranging from 7-49, with higher scores indicating higher experiential avoidance)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean AAQ-II Score (Pre-Intervention) | 27.38 (1.37) | 25.38 (1.43)
  Mean AAQ-II Score (Post-Intervention) | 24.32 (1.40) | 20.93 (1.47)
  Mean AAQ-II Score (1 Month Follow Up) | 23.08 (1.41) | 22.02 (1.47)

48. Other Pre Specified Outcome: Change in Global Distress Tolerance
Description: Distress Tolerance Scale (a 15-item scale ranging from 1-5, with higher scores indicating higher distress tolerance)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean DTS Score (Pre-Intervention) | 3.16 (0.13) | 3.30 (0.14)
  Mean DTS Score (Post-Intervention) | 3.50 (0.14) | 3.61 (0.14)
  Mean DTS Score (1 Month Follow Up) | 3.49 (0.14) | 3.67 (0.15)

49. Other Pre Specified Outcome: Change in Global Self-Compassion
Description: Self-Compassion Scale (a 25-item scale ranging from 1-5, with higher scores indicating higher self-compassion)
Time Frame: as for outcome 11
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness | Coping
Number analyzed (Participants) | 42 | 39
score on a scale
  Mean SCS Score (Pre-Intervention) | 2.63 (0.11) | 2.84 (0.11)
  Mean SCS Score (Post-Intervention) | 2.97 (0.12) | 3.20 (0.12)
  Mean SCS Score (1 Month Follow Up) | 3.17 (0.13) | 3.26 (0.13)

ADVERSE EVENTS:
Time Frame: 8 Weeks
Arm/Group | Mindfulness | Coping
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/39
Other Adverse Events (participants affected / at risk) | 0/42 | 0/39

LIMITATIONS AND CAVEATS:
Seven participants who met initial abbreviated CTQ inclusion thresholds on the online prescreening, but not full CTQ inclusion thresholds at the pre-intervention study visit, were enrolled before a coding error was discovered that flagged participants with scores one point below the CTQ threshold as eligible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT05516108/Prot_SAP_001.pdf
  • Informed Consent Form (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT05516108/ICF_000.pdf